CLINICAL TRIAL: NCT01392417
Title: Anterior Prolift Versus Posterior Prolift for Pelvic Floor Prolapse
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, menahem neuman, Principal Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: 920090043
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2011-07

CONDITIONS: Pelvic Floor Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Women who had surgery for pelvic floor prolapse underwent surgery by anterior Prolift or Posterior prolift at least a year after the surgery.

The data from the charts and from telephone conversations with the patients will be entered to a database. Physical examination data will also be incorporated.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent surgery by anterior Prolift or posterior Prolift for pelvic floor prolapse

Exclusion Criteria:

* Women who did not have surgery by Prolift for pelvic floor prolapse

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic floor prolapse who underwent surgery with Prolift
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of pelvic floor prolapse | One year after surgery
  We will question the women if they have a feeling of a mass protruding through the labia. Physical examination data will also be incorporated.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Obstetrics and Gynecology, Western Galilee Hospital, Nahariya
  - Clinics of Dr Neuman, Tel Aviv